CLINICAL TRIAL: NCT00391976
Title: The Microbiologic Efficacy and Safety of Two Treatment Regimens of Inhaled Tobramycin Nebuliser Solution (TNS) for the Treatment of Early Onset Pseudomonas Aeruginosa Lower Respiratory Tract Infection in Subjects With Cystic Fibrosis
Brief Title: Efficacy and Safety of 28 or 56 Day Treatment for Pseudomonas Aeruginosa in Children With Cystic Fibrosis
Acronym: ELITE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTBM100B2301
Record Dates: First submitted 2006-10-19; First posted 2006-10-25 (Estimated); Results first posted 2011-08-29 (Estimated); Last update posted 2011-08-29 (Estimated); Status verified 2011-07

CONDITIONS: Cystic Fibrosis
Keywords: Cystic fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — Inhalation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tobramycin 300 mg for 28 days (Experimental): Patients inhaled tobramycin 300 mg bis in die (bid, twice a day) for 28 days using the PARI LC PLUS™ jet nebulizer and a suitable compressor. The 2 daily doses were taken approximately 12 hours apart and no less than 6 hours apart.
  Interventions: Drug: Tobramycin solution for inhalation 300 mg
- Tobramycin 300 mg for 56 days (Experimental): Patients inhaled tobramycin 300 mg bis in die (bid, twice a day) for 56 days using the PARI LC PLUS™ jet nebulizer and a suitable compressor. The 2 daily doses were taken approximately 12 hours apart and no less than 6 hours apart.
  Interventions: Drug: Tobramycin solution for inhalation 300 mg

INTERVENTIONS:
Drug: Tobramycin solution for inhalation 300 mg — Tobramycin solution for inhalation was supplied in 5 mL liquid-filled low-density polyethylene ampoules containing 300 mg tobramycin. Patients used a nebulizer to inhale the contents of the ampoules.

SUMMARY:
This study assessed time to recurrence of infection with Pseudomonas aeruginosa following treatment of the initial infection with tobramycin nebuliser solution. The safety profile of the initial tobramycin treatment was assessed during the first 3 months of the study and patients were followed until the end of the study, month 27.

DETAILED DESCRIPTION:
This was a multi-center, open-label, two-arm, randomized study. All patients diagnosed with CF and who fulfilled the criteria for early infection with P. aeruginosa initially received tobramycin 300 mg twice a day for 28 days. At the end of the 28-day treatment period, patients who met the inclusion criteria and none of the additional exclusion criteria were randomized in a 1:1 ratio to either receive an additional 28 days of treatment with tobramycin 300 mg twice a day (56-day group) or to stop study medication (28-day group).

All randomized patients had regular study visits until a positive P. aeruginosa sample was obtained. Once P. aeruginosa had recurred, the patient entered a follow-up phase where minimal information was collected for 27 months. During the follow-up phase, patients were treated according to their physicians' discretion.

Patients who started treatment with tobramycin but were not randomized (i.e. due to a positive antibody test) and followed up during routine clinic visits. They were allowed to continue their 28-day treatment period and afterwards be treated according to their physicians' discretion.

ELIGIBILITY:
Inclusion criteria:

* Male or female patients ≥ 6 months old
* Diagnosis of cystic fibrosis (CF) based upon the following historical criteria performed prior to study participation:

  1. confirmed sweat chloride > 60 mEq/L by quantitative pilocarpine iontophoresis (at least 2 tests), OR
  2. genotype with two identifiable mutations consistent with CF.
* First or early lower respiratory tract infection with Pseudomonas (P.) aeruginosa documented by either of the following:

  1. first infection defined by the first P. aeruginosa isolated from sputum or deep throat cough swab culture, OR
  2. P. aeruginosa from sputum or deep throat cough swab culture following at least 1 year of negative cultures (documented with at least 4 negative cultures during this year and no positive cultures) and no anti-pseudomonal treatment during this 1-year period, OR
  3. P. aeruginosa from sputum or deep throat cough swab culture following at least 2 years of negative cultures (documented with at least 2 negative cultures per year and no positive cultures) and no anti-pseudomonal treatment during this 2-year period.
* Written informed consent by the patient and/or parent/legal guardian according to local country regulations.

Exclusion criteria:

* History of aminoglycoside hypersensitivity or adverse reaction to inhaled aminoglycoside.
* Signs and symptoms of acute pulmonary disease, eg, pneumonia, pneumothorax.
* Administration of any investigational drug within 30 days prior to enrollment.
* Administration of loop diuretics within 7 days prior to study drug administration.
* Personal/family history of abnormal hearing, other than typical hearing loss associated with the aging process.
* Abnormal result from an audiology testing (defined as either a unilateral pure-tone audiometry test showing a threshold elevation > 20 decibels [dB] at any frequency across the frequency range 0.25-8 kHz or the absence of emission at the evoked otoacoustic emission test).
* Positive urine pregnancy test at Day 1 (Baseline) for all female patients who have reached menarche.
* Use of macrolide antibiotics as a maintenance therapy for 12 or more days during the 28 days prior to Baseline.
* Antibody titers ≥ 1000 for any of the 3 P. aeruginosa exoenzymes: Exotoxin A, alkaline protease, or elastase (status to be determined between Baseline and Day 28).

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2003-11; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Felix Ratjen, Principal Investigator — Royal Victoria Infirmary

REFERENCES:
- [Derived] Ratjen F, Munck A, Kho P, Angyalosi G; ELITE Study Group. Treatment of early Pseudomonas aeruginosa infection in patients with cystic fibrosis: the ELITE trial. Thorax. 2010 Apr;65(4):286-91. doi: 10.1136/thx.2009.121657. Epub 2009 Dec 8. PMID 19996339

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 123 patients were enrolled and received tobramycin 300 mg twice a day for 28 days. Patients who received treatment but tested positive for antibodies to any of 3 Pseudomonas aeruginosa exoenzymes in a blood sample collected at baseline were not randomized into one of the two treatment groups but were followed-up during routine clinic visits.
Groups:
- Tobramycin 300 mg for 28 Days: Patients inhaled tobramycin 300 mg twice a day for 28 days using the PARI LC PLUS™ jet nebulizer and a suitable compressor. The 2 daily doses were taken approximately 12 hours apart and no less than 6 hours apart.
- Tobramycin 300 mg for 56 Days: Patients inhaled tobramycin 300 mg twice a day for 56 days using the PARI LC PLUS™ jet nebulizer and a suitable compressor. The 2 daily doses were taken approximately 12 hours apart and no less than 6 hours apart.
- Non-randomized Patients: Patients who started the study and received tobramycin 300 mg twice a day for 28 days, but tested positive for antibodies to any of 3 Pseudomonas aeruginosa exoenzymes in a blood sample collected at baseline were not randomized into the treatment groups. These patients were not included in the efficacy analyses.
Period: Overall Study
Arm/Group | Tobramycin 300 mg for 28 Days | Tobramycin 300 mg for 56 Days | Non-randomized Patients
Started | 45 (Started indicates all patients who were enrolled at Visit 1) | 43 | 35
Randomized | 45 (Randomization occurred after 28 days of treatment & negative antibody test aeruginosa antibody test) | 43 | 0
Safety Population | 44 (Patients who were enrolled and received at least one dose of study medication.) | 43 | 35
Completed | 18 | 18 | 0
Not Completed | 27 | 25 | 35
Not completed — Adverse Event | 0 | 0 | 1
Not completed — Withdrawal of consent | 0 | 1 | 1
Not completed — Lost to Follow-up | 1 | 2 | 0
Not completed — Inappropriate enrollment | 1 | 1 | 0
Not completed — Protocol deviation/violation | 4 | 2 | 1
Not completed — Recurrence/no eradication of infection | 21 | 19 | 0
Not completed — Unable to classify | 0 | 0 | 1
Not completed — Positive P. aeruginosa antibody test | 0 | 0 | 31

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tobramycin 300 mg for 28 Days | Tobramycin 300 mg for 56 Days | Non-randomized Patients | Total
Number analyzed (Participants) | 45 | 43 | 35 | 123
Age Continuous [Mean (Standard Deviation); unit: years] | 8.70 (7.22) | 8.65 (10.54) | 9.09 (5.76) | 8.79 (8.14)
Age, Customized [Number; unit: participants]
  6 months - < 6 years | 19 | 18 | 11 | 48
  6 years - < 18 years | 20 | 21 | 21 | 62
  ≥ 18 years | 6 | 4 | 3 | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 21 | 19 | 59
  Male | 26 | 22 | 16 | 64

OUTCOME MEASURES:

1. Primary Outcome: Time to Recurrence of Pseudomonas (P.) Aeruginosa (Any Genotype) in Sputum or Deep Throat Cough Swab
Description: Microbiological samples were obtained from sputum or by deep throat cough swab technique. Time to recurrence was defined as the time between the visit at 1 month after the end of treatment (when eradication was confirmed) and the time of the first positive culture with any genotype of P. aeruginosa. Time zero was Day 56 (Month 2) for the 28-day treatment group and Month 3 for the 56-day treatment group. Kaplan-Meier estimates were used.
Time Frame: From 1 month after the end of treatment (Day 56 for the 28-day treatment group and Month 3 for the 56-day treatment group) until the end of the study (Month 27)
Population: Efficacy evaluable population: All randomized patients who had microbiological assessments 1 month after their last dose of study drug, except for patients with no eradication 1 month after the last dose of study drug, low compliance (> 50% of capsules returned unused), or violation of protocol procedure in relation to the efficacy analysis.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Non-randomized: Patients who started the study and received tobramycin 300 mg twice a day for 28 days, but tested positive for antibodies to any of 3 Pseudomonas aeruginosa exoenzymes in a blood sample collected at baseline were not randomized into the treatment groups. These patients were not included in the efficacy analyses.
Arm/Group | Tobramycin 300 mg for 28 Days | Tobramycin 300 mg for 56 Days | Non-randomized
Number analyzed (Participants) | 34 | 31 | 0
Months | 26.12 [14.69 to NA] — An upper limit for the CI could not be estimated because of insufficient number of events. | 25.82 [18.17 to NA] — An upper limit for the CI could not be estimated because of insufficient number of events. |

2. Secondary Outcome: Percentage of Patients With Pseudomonas (P.) Aeruginosa Eradicated From Deep Throat Cough Swab or Sputum
Description: One month after the end of treatment was Day 56 (Month 2) for the 28-day treatment group and Month 3 for the 56-day treatment group.
Time Frame: From 1 month after the end of treatment until the end of the study (Month 27)
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Tobramycin 300 mg for 28 Days | Tobramycin 300 mg for 56 Days | Non-randomized
Number analyzed (Participants) | 34 | 31 | 0
Percentage of participants
  At 1 month after the end of treatment | 100 | 100 |
  At final visit | 68 | 71 |

3. Secondary Outcome: Time to Recurrence of Pseudomonas (P.) Aeruginosa (New or Same Genotype) in Sputum or Deep Throat Cough Swab Based on Confirmatory Assessment by the Central Laboratory
Description: Time to recurrence was defined as the time between the visit at 1 month after the end of treatment (when eradication was confirmed) and the time of the first positive culture with any genotype of P. aeruginosa. Time zero was Day 56 (Month 2) for the 28-day treatment group and Month 3 for the 56-day treatment group.
Time Frame: From 1 month after the end of treatment until the end of the study (Month 27)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Tobramycin 300 mg for 28 Days | Tobramycin 300 mg for 56 Days | Non-randomized
Number analyzed (Participants) | 14 | 7 | 0
Months | 9.84 (2.47) [2.73 to 22.57] | 16.62 (2.61) [6.41 to 18.17] |

4. Secondary Outcome: Percentage of Patients With Pseudomonas (P.) Aeruginosa Having an Increased, Decreased, or Unchanged Tobramycin Minimum Inhibitory Concentration (MIC) Value at the Final Visit Compared to Baseline
Description: The percentage of patients with changes in tobramycin MIC values from Baseline to the final visit could not be compared as there was insufficient data.
Time Frame: From Baseline to the final visit (end of the study, Month 27)
Population: Safety population: All patients who were enrolled in the study and received at least 1 dose of study medication.
Measure: Number; unit: Percentage of participants
Arm/Group | Tobramycin 300 mg for 28 Days | Tobramycin 300 mg for 56 Days | Non-randomized
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: Number of Participants Hospitalized for Pulmonary Exacerbations
Description: Core study defined as from Baseline through to one month after the end of treatment (Day 56 for the 28-day treatment group and Month 3 for the 56-day treatment group). Follow-up phase began at the end of the core study through to the end of the study (Month 27).
Time Frame: From Baseline to end of study (27 months)
Population: All patients who were randomized and received at least one dose of study medication. Non-randomized patients were not included in the analysis.
Measure: Number; unit: Participants
Arm/Group | Tobramycin 300 mg for 28 Days | Tobramycin 300 mg for 56 Days | Non-randomized
Number analyzed (Participants) | 44 | 43 | 0
Participants
  Core Study | 0 | 2 (9.2) |
  Follow-up | 5 | 2 |

ADVERSE EVENTS:
Time Frame: From Baseline to the end of the study (Month 27)
Description: Adverse events (AE) were recorded for the safety population which included all patients who received at least 1 dose of study medication. For patients withdrawn from the study who continued in the follow-up phase, all AEs were recorded until Month 3. After Month 3, only AEs recorded related to study drug were recorded.
Groups:
- Tobramycin 28 Days Up To Month 3: Patients inhaled tobramycin 300 mg twice a day for 28 days using the PARI LC PLUS™ jet nebulizer and a suitable compressor. The 2 daily doses were taken approximately 12 hours apart and no less than 6 hours apart.
- Tobramycin 56 Days Up To Month 3: Patients inhaled tobramycin 300 mg twice a day for 56 days using the PARI LC PLUS™ jet nebulizer and a suitable compressor. The 2 daily doses were taken approximately 12 hours apart and no less than 6 hours apart.
- Non-randomized Patients up to Month 3: Patients who started the study and received tobramycin 300 mg twice a day for 28 days but tested positive for antibodies to any of 3 Pseudomonas aeruginosa exoenzymes in a blood sample collected at baseline were not randomized into the treatment groups.
- Tobramycin 28 Days After Month 3: Patients who received tobramycin 300 mg twice a day for 28 days using the PARI LC PLUS™ jet nebulizer and a suitable compressor. Patients received no study medication during the follow-up phase (from Month 3 though Month 27).
- Tobramycin 56 Days After Month 3: Patients received tobramycin 300 mg twice a day for 56 days using the PARI LC PLUS™ jet nebulizer and a suitable compressor. Patients received no study medication during the follow-up phase (from Month 3 though Month 27).
Arm/Group | Tobramycin 28 Days Up To Month 3 | Tobramycin 56 Days Up To Month 3 | Non-randomized Patients up to Month 3 | Tobramycin 28 Days After Month 3 | Tobramycin 56 Days After Month 3
Serious Adverse Events (participants affected / at risk) | 4/44 | 3/43 | 1/35 | 2/35 | 2/36
Other Adverse Events (participants affected / at risk) | 23/44 | 14/43 | 3/35 | 19/35 | 18/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tobramycin 28 Days Up To Month 3 (N=44) | Tobramycin 56 Days Up To Month 3 (N=43) | Non-randomized Patients up to Month 3 (N=35) | Tobramycin 28 Days After Month 3 (N=35) | Tobramycin 56 Days After Month 3 (N=36)
CONSTIPATION (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
PYREXIA (General disorders) | 0 | 0 | 0 | 0 | 1
BRAIN ABSCESS (Infections and infestations) | 0 | 0 | 0 | 1 | 0
GASTROENTERITIS (Infections and infestations) | 0 | 1 | 0 | 0 | 0
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 0 | 1 | 0 | 0
OTITIS MEDIA (Infections and infestations) | 0 | 0 | 0 | 1 | 0
PSEUDOMONAS INFECTION (Infections and infestations) | 2 | 0 | 0 | 0 | 0
STENOTROPHOMONAS INFECTION (Infections and infestations) | 1 | 0 | 0 | 0 | 0
VARICELLA (Infections and infestations) | 0 | 1 | 0 | 0 | 0
GRAND MAL CONVULSION (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
DYSPHONIA (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
HYDROCELE OPERATION (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tobramycin 28 Days Up To Month 3 (N=44) | Tobramycin 56 Days Up To Month 3 (N=43) | Non-randomized Patients up to Month 3 (N=35) | Tobramycin 28 Days After Month 3 (N=35) | Tobramycin 56 Days After Month 3 (N=36)
VOMITING (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 3
PYREXIA (General disorders) | 3 | 4 | 0 | 2 | 1
BRONCHITIS (Infections and infestations) | 2 | 0 | 0 | 3 | 4
NASOPHARYNGITIS (Infections and infestations) | 3 | 0 | 0 | 0 | 2
OTITIS MEDIA (Infections and infestations) | 0 | 1 | 0 | 2 | 2
RHINITIS (Infections and infestations) | 7 | 3 | 1 | 3 | 2
SINUSITIS (Infections and infestations) | 0 | 0 | 0 | 2 | 0
TONSILLITIS (Infections and infestations) | 1 | 0 | 0 | 4 | 1
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 4 | 2 | 0 | 4 | 4
VARICELLA (Infections and infestations) | 0 | 0 | 0 | 0 | 3
HEADACHE (Nervous system disorders) | 3 | 1 | 0 | 0 | 0
COUGH (Respiratory, thoracic and mediastinal disorders) | 9 | 2 | 1 | 9 | 7
DYSPHONIA (Respiratory, thoracic and mediastinal disorders) | 5 | 5 | 1 | 0 | 0
LUNG DISORDER (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 1 | 2
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.